CLINICAL TRIAL: NCT02634632
Title: Assessments and Recommendations for the Implementation of Advance Directives in Oncology
Acronym: DA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-22; 2015-A00692-47 (Registry Identifier: ID RCB); RCAPHM15_0141 (Other: AP-HM)
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Patient Having a Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with cancer (Experimental): choose to write advance directives
  Interventions: Behavioral: Choosing to write advance directives

INTERVENTIONS:
Behavioral: Choosing to write advance directives

SUMMARY:
Legitimized by the Leonetti law of April 22, 2005, advance directives (AD) appear in various places of care that alongside the end of life, and even tend to be generalized to all areas related to health care in general. In this context, a prospective study to assess how the patient will seize the AD and identify the different problems writing these AD will be conducted. From this study, it will establish recommendations for the implementation of AD in the Multidisciplinary Oncology Department and Therapeutic Innovations service and in oncology in general. They will be asked patients if they choose to write their AD, complete and sign the AD pre-written in the book or not to draft their AD. The choice of the patients, but also the reasons they associate thereto and, where appropriate, their AD written will be collected. The patient will also inform its demographic and socio the case report (clinical data) should be completed by the investigator. During the first part of research, the use of AD by patients and will be assessed and analyzed in connection with the characteristics of these patients (history of the disease, course of care, socio-demographic) and the reasons they set out to explain their choice. For those who write their AD, they will, in a second step, subject to thematic content analysis to identify the main aspects that the subject convened to consider its end of life.This research therefore lead to the definition of the contours of a user device AD in oncology in general. This study was qualified biomedical research because of the sensitive nature of the study population and bring the patient to personal preoccupations when filling the questionnaire on the choice of directing advance directives and their contents.

ELIGIBILITY:
Inclusion Criteria:

* Subject both sexes
* Subject whose age is between 18 and 85 years
* Subject with cancer
* Subjects for which French is the native language, about having read, understood and signed the informed consent

Exclusion Criteria:

* Subject minors or subjects aged over 85 years
* Subject not including the French
* Subject with neurological or psychiatric disorders prohibiting their understanding of the study
* Subject private freedom following a judicial or administrative decision

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation the rate of use of advance directives | 24 months
  survey

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France